CLINICAL TRIAL: NCT03573258
Title: Effects of Dietary Fibre on Satiety in Morbidly Obese Patients Before and After Bariatric Surgery - a Single Center, Randomized, Single-blinded, Cross-over Study.
Brief Title: Dietary Fibers and Satiety in Bariatric Patients
Acronym: FIBAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Marco Bueter, Prof. Dr. med., PhD, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ID 2017-02287
Record Dates: First submitted 2018-04-20; First posted 2018-06-29 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded cross-over trial in 24 morbidly obese human subjects undergoing RYGB.
Who Masked: Participant
Masking Description: single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber (Experimental): 300 ml of orange juice plus Intervention
  * 6 g of oat beta glucan = FIBER (study A) or
  * 25 g inulin/FOS = FIBER (study B)
  Interventions: Dietary Supplement: Fiber or Placebo (depending on the randomization)
- Placebo (Placebo Comparator): 300 ml of orange juice plus Placebo:
  * 13.5 g maltodextrin = PLACEBO (study A) or
  * 15.5 g maltodextrin = PLACEBO (study B)
  Interventions: Dietary Supplement: Fiber or Placebo (depending on the randomization)

INTERVENTIONS:
Dietary Supplement: Fiber or Placebo (depending on the randomization) — ingestion of dietary fibers prior to meal intake
  Other Names: Placebo

SUMMARY:
The primary objective is to evaluate the effect of a viscous and fermentable dietary fibre on ad libitum eating in morbidly obese patients before and 6 month after Roux-en-Y gastric bypass (RYGB) surgery.

The secondary objectives are to study the effect of a viscous and fermentable dietary fibre on perceived appetite, the production of short chain fatty acids (SCFA), breath hydrogen (as a marker of large intestinal fermentation), the secretion of gastrointestinal (GI) satiation hormones and glycaemia in morbidly obese patients before and 6 month after RYGB surgery.

The primary study outcome measure is macronutrient and food intake (grams and kcal eaten) at the ad libitum buffet meal as well as time to complete the meal.

Secondary outcome measures are 1) Appetite ratings (validated visual analogue scales, VAS) including hunger, fullness, thirst, desire to eat, and amount of food desired to eat. 2) Plasma concentrations of SCFA (propionate, acetate, butyrate). 3) Breath hydrogen (as a marker of large intestinal fermentation) 4) Plasma concentrations of gastrointestinal hormones (ghrelin, cholecystokinin (CCK), glucagon-like peptide-1 (GLP-1), peptide YY (PYY) and potentially other, yet to be identified gut hormones). 4) Concentrations of plasma insulin and glucagon and blood glucose.

Randomized, single-blinded cross-over trial in 24 morbidly obese human subjects undergoing RYGB (study A, n=12; study B, n=12). Study B also includes an additional pilot study in 6 morbidly obese patients before and 6 month after RYGB surgery. Thus, the total number of subjects including the pilot study is 30.

DETAILED DESCRIPTION:
Obesity has reached epidemic proportions worldwide. The only effective treatment option currently available is bariatric surgery, with the gold standard procedure, the Roux-en-Y gastric bypass (RYGB), resulting in dramatic and sustained excess weight loss of 60-75% and often prompt amelioration of type 2 diabetes mellitus (T2DM). The unparalleled efficacy of bariatric surgery in obesity treatment opens a completely new perspective for the development of anti-obesity drugs, and suggests that the gastrointestinal (GI) tract is of much more importance in the control of eating and energy homeostasis than previously thought.Two key GI mechanisms have been identified to inhibit eating: 1) gastric distention resulting in activation of mechanoreceptors and neural gut brain signaling, and 2) small intestinal nutrient sensing resulting in the secretion of satiation peptides such as CCK, GLP-1 and PYY.

A completely novel implication of the importance of the GI tract in the control of eating and body weight is the role of the large intestine and the gut microbiome as well as its metabolic products.That the gut microbiome can have potent effects on eating and body weight was first recognized in landmark experiments with germ-free mice that became obese when they were inoculated with microbiota from obese mice or humans, while they remained lean when microbiota was transplanted from lean mice.

The exact mechanisms that link the gut microbiome to the control of eating and energy homeostasis remain however, largely unexplored. One suggestion for obesity development is that the 'obese' microbiome may have an increased capacity to extract energy from the same diet as compared with a 'lean' microbiome. In fact, short chain fatty acids (SCFA) formed through bacterial fermentation of indigestible carbohydrates can provide additional energy to the host (about 10% of total energy from the diet). However, whether this is the main cause for obesity development remains controversial because SCFA also stimulate the secretion of leptin, GLP-1 and PYY and, thus, activate eating-inhibitory mechanisms. Because under physiological conditions, a meal will take about 6 hours or longer (depending on meal composition and inter-individual variability of intestinal transit) until it reaches the large intestine so that fermentable meal components can be metabolized to SCFA, the contribution of SCFA in acute eating-inhibitory effects has been questioned in humans. Bariatric patients provide an ideal model to study this mechanism. Based on the anatomical alterations during RYGB surgery resulting in a much faster nutrient transit to the large intestine, it can be hypothesized that a more rapid and more pronounced production of SCFA contributes to the marked acute eating-inhibitory effects as seen after surgery. In addition, RYGB patients have a small stomach pouch about 2% of the size of a normal, un-operated stomach resulting in early distention upon food ingestion. The effect of increased stomach distention and its contribution to the overall effects on eating behavior and weight loss have not been evaluated, to the best of our knowledge. Dietary fibres provide an ideal nutritional intervention to study the underlying eating-inhibitory effects of RYGB surgery. 1) High viscous fibres such as oat beta glucan delay gastric emptying and, thus, may contribute to the eating effect via an increase in gastric distention. 2) Non-viscous, fermentable fibres such as inulin or fructo-oligossachides (FOS) are highly fermented into SCFA in the large intestine upon ingestion, and thus may participate in the eating effect via activation of SCFA receptors and release of satiation hormones.

The primary objective in both study A and B is to evaluate the effect of a viscous and fermentable dietary fibre on ad libitum eating in morbidly obese patients before and 6 month after RYGB surgery.

In addition, in the pilot study in study B, the primary objective is the time course of fibre-induced large intestinal fermentation.

The secondary objectives in both study A and B are to study the effect of a viscous and fermentable dietary fibre on perceived appetite, the production of SCFA, breath hydrogen (as a marker of large intestinal fermentation), the secretion GI satiation hormones and glycaemia in morbidly obese patients before and 6 month after RYGB surgery.

The primary study outcome measure in both study A and B is macronutrient and food intake (grams and kcal eaten) at the ad libitum buffet meal as well as time to complete the meal.

In addition, in the pilot study in study B, the primary study outcome measure is breath hydrogen and plasma SCFA concentrations.

Secondary outcome measures in both study A and B are 1) Appetite ratings (validated visual analogue scales, VAS) including hunger, fullness, thirst, desire to eat, and amount of food desired to eat. 2) Plasma concentrations of SCFA (propionate, acetate, butyrate). 3) Breath hydrogen (as a marker of large intestinal fermentation) 4) Plasma concentrations of gastrointestinal hormones (ghrelin, CCK, GLP-1, PYY and potentially other, yet to be identified gut hormones). 4) Concentrations of plasma insulin and glucagon and blood glucose.

Randomized, single-blinded cross-over trial in 24 morbidly obese human subjects undergoing RYGB (study A, n=12; study B, n=12). Study B also includes an additional pilot study in 6 morbidly obese patients before and 6 month after RYGB surgery. Thus, the total number of subjects including the pilot study is 30.

ELIGIBILITY:
Inclusion criteria:

* Morbidly obese patients undergoing RYGB surgery
* Male or female, age 18 or over
* Sufficient understanding of the German language
* Understand the procedures and the risks associated with the study
* Willing to adhere to the protocol and sign the consent form (dietary/physical restrictions are a) no alcohol and no xanthine-containing liquids such as coffee, black or green tea, cola, red bull, chocolate 24 h before the study sessions. b) an identical dinner the evening before the study sessions followed by fasting overnight with no additional food or fluid except water. c) no strenuous exercise for 24 h before each treatment)
* Independently mobile

Exclusion Criteria:

* Pregnancy or lactation (as determined by questionnaire and/or pregnancy test)
* Active and significant psychiatric illness including substance misuse
* Significant cognitive or communication issues
* Medications with documented effect on food intake or food preference
* History of significant food allergy and certain dietary restrictions (e.g. Lactose intolerance)
* Participation in another clinical trial (currently or within the last 30 days)
* Smoking
* Chronic or acute medical condition including clinically relevant abnormality in physical exam or laboratory values
* Consumption of high fiber diets (e.g. vegans, etc.) or fiber supplements or pre and probiotics
* Pre-operatively: Factors impairing ability to consume a meal such as significant dysphagia, gastric outlet obstruction, or any other factor that prevents subjects from drinking or eating a meal
* Post-operatively: Factors impairing the ability to consume meal such as significant and persistent surgical complications, any other factors that prevents subjects from drinking or eating a meal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
food intake | 75 (study A) /180 (study B) minutes after Fiber intake
  macronutrient and food intake (grams and kcal eaten) at the ad libitum buffet meal
fermentation | up to 5 hours after fiber intake
  breath hydrogen

SECONDARY OUTCOMES:
Appetite ratings on hunger, fullness and satiety | up to 5 hours after fiber intake
  100 mm visual analogue scales (range 0 to 100, representing the strenght of the feeling)
short chain fatty acid levels | 150 (study A) / 270 (study B) minutes after Fiber intake
  Plasma concentrations of SCFA (propionate, acetate, butyrate)
gut hormones | 150 (study A) / 270 (study B) minutes after Fiber intake
  Plasma concentrations of gastrointestinal hormones (ghrelin, CCK, GLP-1, PYY )
glucose metabolism | 150 (study A) / 270 (study B) minutes after Fiber intake
  Concentrations of plasma insulin and glucagon and blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bueter, MD PhD, Principal Investigator — University Hsopital Zurich, Visceral Surgery
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Information about study subjects will be kept confidential and managed according to the Cantonal Ethical requirements. Access to any information that could link study data to individual subjects will be strictly limited to research personnel involved in the study and the study monitor. Any data forms that include identifying information will be kept in locked files at the University Hospital Zurich (USZ). Data will be recorded on case report forms. Any reports, scientific papers or presentations will not include any information that could be used to identify individuals.

REFERENCES:
- [Background] Slavin J. Fiber and prebiotics: mechanisms and health benefits. Nutrients. 2013 Apr 22;5(4):1417-35. doi: 10.3390/nu5041417. PMID 23609775
- [Background] Clark MJ, Slavin JL. The effect of fiber on satiety and food intake: a systematic review. J Am Coll Nutr. 2013;32(3):200-11. doi: 10.1080/07315724.2013.791194. PMID 23885994